CLINICAL TRIAL: NCT07171125
Title: Liposomal Bupivacaine for Acute Pain Management Following Posterior Lumbar Decompression and Fusion Surgery in Adults: A Prospective, Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine for Pain After Lumbar Fusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Min Li (Other)
Responsible Party: Sponsor-Investigator, Min Li, Professor and Chief Physician, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M20250040
Record Dates: First submitted 2025-08-27; First posted 2025-09-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Acute Pain; Lumbar Degenerative Diseases
Keywords: Liposomal bupivacaine; Local infiltration analgesia; Posterior lumbar fusion; Postoperative pain; Randomized controlled trial; Opioid-sparing
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All personnel responsible for short-term and long-term postoperative follow-up, completion of clinical observation forms, and data entry/verification are excluded from patient recruitment, randomization, and anesthesia management. These personnel remain blinded to patient group allocation and are prohibited from communicating with the study coordinator regarding any group assignment information.Statistical analysis is performed by dedicated statisticians not involved in clinical anesthesia procedures.Both patients and their family members remain blinded to group allocation throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine Group (Experimental): 266 mg liposomal bupivacaine + 25 mg bupivacaine HCl, local infiltration during closure
  Interventions: Drug: Liposomal bupivacaine (local infiltration)
- Ropivacaine Group (Active Comparator): 120 mg ropivacaine, local infiltration during closure.
  Interventions: Drug: ropivacaine (local infiltration)

INTERVENTIONS:
Drug: Liposomal bupivacaine (local infiltration) — Patients will receive a pre-closure local infiltration of 266 mg liposomal bupivacaine (20 mL for single-level surgery; 30 mL for two-level surgery) combined with 25 mg bupivacaine hydrochloride (10 mL total volume). The drug will be injected bilateral into the paraspinal muscles and subcutaneous tissues prior to wound closure. This provides both immediate (bupivacaine HCl) and prolonged (liposomal) analgesia."
  Arms: Liposomal Bupivacaine Group
Drug: ropivacaine (local infiltration) — Patients will receive 120 mg ropivacaine diluted to 30 mL (single-level) or 40 mL (two-level) with normal saline. The solution will be infiltrated bilateral into the paraspinal muscles and subcutaneous tissues using the same technique as the experimental arm, ensuring consistent injection depth and distribution.
  Arms: Ropivacaine Group

SUMMARY:
Spine surgery often causes severe postoperative pain. Currently, our hospital routinely uses ropivacaine for local infiltration analgesia (lasting 6-8 hours). This study evaluates liposomal bupivacaine, a novel long-acting local anesthetic providing up to 72 hours of pain relief, in patients undergoing posterior lumbar spine surgery. Through a randomized controlled design, we will compare the two drugs' effects on pain control within 72 hours and opioid consumption. Both regimens are guideline-recommended and safe.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years；
* ASA physical status class I-III；
* Scheduled for elective 1- or 2-level posterior lumbar surgery: Decompression (laminectomy/discectomy) and fusion with internal fixation

Exclusion Criteria:

* Chronic pain disorders requiring ≥30 mg oral morphine equivalents/day for >3 months.
* Pre-existing neurological deficits that may interfere with pain assessment.
* Hypersensitivity to any component of multimodal analgesia or local anesthetics (e.g., bupivacaine, ropivacaine).
* Acute systemic/local infection (e.g., surgical site infection, sepsis).
* Metastatic spinal malignancies (confirmed by imaging/histopathology).
* Pregnancy or lactation.
* Patient refusal after detailed protocol explanation.
* Other investigator-determined high-risk conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption within 72 hours postoperatively (converted to morphine milligram equivalents, MME) | 72 hours postoperative
  Opioid doses will be converted to MME using the CDC standard conversion table

SECONDARY OUTCOMES:
Postoperative pain intensity assessed by Numeric Rating Scale (NRS, 0-10) at rest and during movement (e.g., coughing/ambulation) at predefined timepoints: pre-PACU discharge, 4h, 8h, 24h, 48h, and 72h after surgery. | Immediately prior to PACU discharge，4 hours, 8 hours, 24 hours, 48 hours, and 72 hours after surgery.
  NRS ranges from 0 (no pain) to 10 (worst imaginable pain). Movement-associated pain will be assessed during standardized activities (e.g., coughing on command or first ambulation).All assessors will be trained to ensure consistent NRS measurement across timepoints.
  Daytime assessments: Performed within ±30 minutes of scheduled timepoints
  Nighttime adjustments:
  Assessments falling between 21:00 (9:00 PM) and 07:00 (7:00 AM) will be deferred to 08:00 AM the following morning to avoid sleep disruption.
  Original timepoints documented with annotations (e.g., "Scheduled: 02:00; Assessed: 08:00+1")
Total postoperative morphine consumption via PCA | Cumulative consumption recorded at 4 hours, 8 hours, 24 hours, 48 hours, and 72 hours after surgery
  PCA settings will be standardized across all patients:
  * Bolus dose: 1 mg morphine equivalent
  * Lockout interval:10 minutes
  * No background infusion.
Total Postoperative Rescue Tramadol Consumption | From PCA initiation until 72 hours (Day3) postoperatively. Rescue tramadol consumption will be recorded at 4hours, 8hour, 24hours, 48hours, 72hours after surgery.
  Trigger Criteria: NRS >3 at rest despite PCA morphine (1mg bolus, 10min lockout).
  Dosing Protocol: Tramadol 50mg IV/oral
  Data Collection:
  Cumulative tramadol consumption recorded at 4hours, 8hour, 24hours, 48hours, 72hours after surgery.
  Convert oral to IV equivalent for analysis
Sleep disturbance due to pain (binary scale) | Postoperative Days 1 (24 hours), 2 (48 hours), and 3 (72 hours), with daily assessment window: 8:00-9:00 AM
  Patients will report whether pain interfered with sleep during the previous night using a standardized binary scale:
  * 0: No sleep disruption (pain did not awaken or prevent sleep)
  * 1: Sleep disrupted (pain caused awakening or difficulty falling asleep).
  Assessment Protocol:
  Evaluated each morning at 8:00 AM by trained research staff Covers sleep quality during the preceding night (20:00-07:59) Delayed assessment for nighttime surgeries: If surgery ends after 18:00, first assessment deferred to 8:00 AM on postoperative Day 1
Time to first independent ambulation | From surgery completion until event occurs, assessed up to 72 hours postoperatively
  Definition: Hours from surgery end to first unassisted walking >5 meters
Immediate local anesthetic-related complications (0-2 hours) | From local anesthetic infiltration completion through 2 hours post-procedure.
  All complications will be recorded and graded. Immediate events (0-2h):
  * Local anesthetic systemic toxicity (LAST): CNS/CV symptoms (e.g., seizures, arrhythmias)
  * Allergic reactions: urticaria, bronchospasm, anaphylaxis
Incidence of nausea/vomiting (PONV) | From surgery completion through 72 hours (Day 3) postoperatively, with interval reporting: 0-24 hours (Day 1), 24-48 hours (Day 2), 48-72 hours (Day 3).
  Graded by severity: 1=Mild (no rescue), 2=Moderate (required 1 antiemetic), 3=Severe (≥2 antiemetics or prolonged NPO).
  Standardized Assessment Protocol at fixed timepoints:
  Day 1: 0-24 hours postoperatively Day 2: 24-48 hours postoperatively Day 3: 48-72 hours postoperatively
  Assessment window:
  Performed daily at 08:00 AM for previous 24-hour period Evening surgeries (end time >18:00): First assessment at 08:00 AM on Day 1
  Symptom tracking:
  Nursing staff document all emetic episodes and antiemetic administrations in real-time
Pruritus severity | From surgery completion through 72 hours (Day 3) postoperatively, with interval analyses: 0-24 hours (Day 1)，24-48 hours (Day 2)，48-72 hours (Day 3)
  Rated by patients: 0=None, 1=Mild (no treatment), 2=Moderate (topical therapy), 3=Severe (systemic treatment).
Incidence of Postoperative Urinary Retention Requiring Catheterization | From surgery completion through 72 hours (Day 3) postoperatively, with planned intervals: 0-24 hours (Day 1), 24-48 hours (Day 2), 48-72 hours (Day 3).
  Definition & Assessment Protocol:
  Diagnostic Criteria: Bladder volume ≥600 mL (ultrasound-confirmed) + inability to void spontaneously.
  Catheterization threshold: Pain (VAS ≥4) with bladder volume ≥600 mL, OR No voiding for 8 hours + bladder volume ≥400 mL.
  Data Collection:
  Event-driven assessments: Triggered by patient-reported symptoms. Maximum observation period: 72 hours (Day 3).
Postoperative Sedation Levels Assessed by Ramsay Scale | From anesthesia emergence until 72 hours postoperatively, at Fixed timepoints: 4 hours, 8 hours, 24 hours, 48 hours and 72 hours after surgery.
  Ramsay Scale:
  1. Patient anxious/agitated
  2. Cooperative/oriented
  3. Responds to commands only
  4. Asleep but brisk response to stimulus
  5. Sluggish response
  6. No response.
  Scoring Direction: Higher scores indicate deeper sedation (1=inadequate, 6=excessive).
  Clinical Thresholds:
  Target range: RSS 2-4 (ERAS-recommended optimal sedation) Intervention triggers: RSS ≥5 (reduce sedation), RSS ≤1 (rescue analgesia)
  Assessment Protocol
  Fixed Timepoints:
  4 hours (Postoperative Day 0) 8 hours (Postoperative Day 0) 24 hours (Postoperative Day 1) 48 hours (Postoperative Day 2) 72 hours (Postoperative Day 3)
  Nighttime Adjustment:
  Assessments between 21:00-07:00 deferred to 08:00 next morning Data Collection Window: ±30 minutes at each timepoint
  Standardized Stimuli:
  Verbal: "Open your eyes" at 70 dB Tactile: Shoulder shaking with 500g pressure
Incidence of Postoperative Delirium Assessed by 3D-CAM (3-Minute Diagnostic Interview for CAM-Defined Delirium) | From anesthesia emergence through 72 hours postoperatively: Primary Assessment Points: 24 hours (Postoperative Day 1) 48 hours (Postoperative Day 2) 72 hours (Postoperative Day 3)
  3D-CAM assesses: 1) Acute onset, 2) Inattention, 3) Disorganized thinking, 4) Altered consciousness. Administered by trained research assistants blinded to group allocation.
  Primary Assessment Points:
  24 hours (Postoperative Day 1) 48 hours (Postoperative Day 2) 72 hours (Postoperative Day 3)
  Evaluation Window:
  ± 30 min at each timepoint. Nighttime detections (21:00-07:00) formally assessed at 08:00 next morning
PCA demand attempts | Counted over consecutive intervals: 0-4 hours, 4-8 hours, 8-24 hours, 24-48 hours, and 48-72 hours postoperatively
  Unit of Measure: Number of attempts
PCA delivery/demand ratio | Calculated for each interval: 0-4hours, 4-8hours, 8-24hours, 24-48hhours, 48-72hours after surgery.
  Calculation: (Number of successful PCA deliveries / Number of PCA demand attempts) × 100
Time to first PCA attempt | Recorded from end of surgery until first PCA button press
Time to first tolerated oral intake | From PACU discharge until event occurs, assessed up to 48 hours postoperatively
  Definition: Hours from surgery end to first clear liquid intake (≥50 mL) without vomiting within 30 minutes
Time to first bowel movement | From surgery completion until event occurs, assessed up to 7 days postoperatively
  Definition: Hours from surgery end to first flatus or defecation reported by patient
Postoperative length of stay | From surgery completion until discharge, assessed up to 14 days postoperatively
  Definition: Days from surgery end to hospital discharge (excluding preoperative days)
Delayed local anesthetic-related complications (24-72 hours) | Any clinical suspicion triggers immediate evaluation from 24 hours (Day 1) through 72 hours (Day 3) postoperatively
  Definition: Complications manifesting 24-72 hours postoperatively
  Subcategories:
  1.Wound Complications:
  1. Infection: CDC criteria (purulent drainage + ≥1: erythema, pain, swelling)
  2. Hematoma: Ultrasound-confirmed collection >5 mL + hemoglobin drop ≥1 g/dL
  3. Neurological Injury 2.Persistent deficit: Sensory/motor dysfunction beyond 72 hours Confirmed by: Day 3: Nerve conduction studies (amplitude reduction >50%). Day 7: EMG if symptoms persist
  Assessment Schedule:
  Fixed timepoints: 24h (Day 1), 48h (Day 2), 72h (Day 3) at 08:00 AM Symptom-driven: Any clinical suspicion triggers immediate evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to local data protection regulations, but anonymized aggregate results will be published.